CLINICAL TRIAL: NCT06312059
Title: Growth Tolerance and Safety Study of Healthy Term Infants Consuming a Goat or Cow Milk Based Infant Formula
Brief Title: Goat or Cow Milk Based Infant Formula GMS
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kendal Nutricare Ltd (Industry)
Collaborators: ObvioHealth (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: KNC-GMS-002
Record Dates: First submitted 2024-01-04; First posted 2024-03-15 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2023-12

CONDITIONS: Growth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: RP Over stickered TP in blank packaging.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Market leader- Competitor Cow Milk based infant formula (Active Comparator): Intervention with Competitor product currently in market- Control.
  Interventions: Other: Advance Infant Formula Powder
- Test product Cow Milk based infant formula (Experimental): Intervention with Test product product - Test arm.
  Interventions: Other: "Kendamil Cow milk test product
- Test product Goat Milk based infant formula (Experimental): Intervention with Test product product - Test arm.
  Interventions: Other: "Kendamil goat milk test product

INTERVENTIONS:
Other: Advance Infant Formula Powder — Sole source infant nutrition for the control arm.
  Arms: Market leader- Competitor Cow Milk based infant formula
Other: "Kendamil Cow milk test product — Sole source infant nutrition for the cow milk test arm.
  Arms: Test product Cow Milk based infant formula
Other: "Kendamil goat milk test product — Sole source infant nutrition for the goat milk test arm.
  Arms: Test product Goat Milk based infant formula

SUMMARY:
This study is a non-inferiority, decentralized, randomized, double-blind, controlled clinical trial evaluating the growth, tolerance, and safety of a goat's-milk test infant formula (Test Formula 1; TF1) and a cow's-milk test infant formula (Test Formula 2; TF2), each compared to a cow's-milk infant formula commercially available in the United States (Control Formula; CF).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy term infants (37 to 42 weeks gestation at birth) from a singleton birth as assessed by the investigator
2. Infants with a birth weight of >2500 g to <4500 g
3. Infants ≤11 days of age at enrollment; birth constitutes Day 0
4. Parent/legal guardian who has previously decided to exclusively feed infant formula and is willing to continue with formula feeding throughout the study

Exclusion Criteria:

A participant who meets any of the following criteria will be excluded from participation in the study:

1. Infant born with medical complications (e.g., neurological, cerebral palsy, etc.)
2. Infant with failure to thrive, fever, any GI tract abnormalities (e.g., short gut, gastroesophageal reflux, etc.), any congenital illness or malformation that may affect infant feeding or normal growth
3. Infant has been treated with prescription medications that in the Investigator's opinion could impact growth, gastrointestinal tolerance and/or development
4. Infant that has received oral or parenteral antibiotics prior to enrollment
5. Infant is taking and parent/legal guardian plans to continue (including over-the-counter medications, such as Mylicon® for gas), home remedies (such as juice for constipation), gastroesophageal reflux medications, herbal preparations, or rehydration fluids that, in the Investigator's opinion, might affect gastrointestinal tolerance. Use of the following are strongly discouraged for the duration of the trial:

   1. Solid foods and juices
   2. Vitamins and/mineral supplements, as the study product provided is nutritionally complete
   3. Pre- and probiotics
6. Infant with family history (biological siblings or parents) of confirmed milk protein allergy (Parent's lactose intolerance is not disqualifying)
7. Parent(s)/Legal guardian(s) intent on feeding non-study formula, breastmilk, juices, or solid food during the study.

Max Age: 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 264 (Estimated)
Dates: Start 2023-12-14 (Actual); Primary Completion 2024-08-15 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
Growth as compared against WHO growth charts | 16 weeks
  Mean daily weight gain for infants fed TF1 and infants fed TF2, each compared to infants fed CF, from baseline through to Week 16

SECONDARY OUTCOMES:
Safety | 16 weeks
  Adverse Events reported over the 16-week study period (+4 days) for all groups

OTHER OUTCOMES:
Tolerability- Monitoring of stool consistency | 16 weeks
  • Stool characteristics (using BITSS) at baseline, and Weeks 2, 4, 8, 12, and 16
Tolerability - fussiness | 16 weeks
  • Formula tolerance (using IGSQ) at baseline, and Weeks 2, 4, 8, 12, and 16
Mean Daily Recumbent Length Gain | 16 weeks
  Change from baseline through to Week 16 for infants fed TF1, infants fed TF2, and infants fed CF in:
  o mean daily recumbent length gain
Mean Daily Head Circumference Gain | 16 weeks
  Change from baseline through to Week 16 for infants fed TF1, infants fed TF2, and infants fed CF in:
  o mean daily head circumference gain

CONTACTS AND LOCATIONS:
Overall Officials: Allan Soo, Principal Investigator — MD, FAPCR ObvioHealth USA, Inc.
Locations (1):
- ObvioHealth USA, Inc., New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Information to be shared with regulatory agencies.